CLINICAL TRIAL: NCT00153621
Title: Prevalence of Proteinuria and Chronic Kidney Disease in Pediatric Patients in the Special Immunology, Burgess, and Nephrology Clinics
Brief Title: Prevalence of Proteinuria and Chronic Kidney Disease in Pediatric HIV-Infected Patients
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Other Study IDs: 3406; NCRR 1K12RR017613-01
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Kidney Failure; AIDS-Associated Nephropathy; HIV Infections
Keywords: Pediatrics; Chronic Kidney Failure; HIV; Acquired Immunodeficiency Syndrome; AIDS-Associated Nephropathy
MeSH Terms: conditions — Kidney Failure, Chronic; AIDS-Associated Nephropathy; HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Among adults with Human Immunodeficiency Virus (HIV) and Acquired Immunodeficiency Syndrome (AIDS), Chronic Kidney Disease (CKD) has previously been reported to occur in approximately 10% of children with HIV-infection. The frequency of CKD, its causes, and its natural history in children and adolescents with HIV-infection have not been systematically studied, particularly in the era of new anti-retroviral medications. The primary aim of this study is to determine the how common pediatric HIV-infected individuals have evidence of persistent proteinuria and CKD.

DETAILED DESCRIPTION:
Human Immunodeficiency Virus-infection has been a significant cause of pediatric morbidity and mortality since it was first identified in the early 1980s. In 1997, HIV became the fourth leading cause of death among children 1 to 4 years of age. As of December 2001, there were 9,074 children under the age of 13 years who have been diagnosed with AIDS in the United States and its territories, and an additional 3,923 children with HIV-infection under the age of 13 years. Human Immunodeficiency Virus-infection and AIDS do not affect children equally in the United States. Whereas whites comprise 61% of the pediatric population, they represent only 15-20% of children with HIV or AIDS. In contrast, African-Americans account for only 14% of the US pediatric population, but they represent 60-65% of children with HIV or AIDS. The prevalence rate of AIDS among African-American children in 2001 was 14 times greater than among white children, and 7 times higher than among Hispanic children.

A variety of renal, electrolyte, and acid-base disturbances have been described in patients with HIV-infection. These abnormalities may be associated with the HIV-infection itself, opportunistic infections, antiviral medications, or unrelated primary disorders. Proteinuria may serve as an early indicator of HIV-associated nephropathy (HIVAN), the pathologic renal lesions associated with HIV-infection itself. Autopsy data in adults with HIV-infection or AIDS have demonstrated a prevalence of HIVAN of between 1 and 15%. The prevalence of HIVAN in the pediatric population has been reported between 7 and 15%. The racial disparity seen in the AIDS population has also been described in the pediatric HIVAN population. Reports of HIVAN in pediatric populations found that 137 of 155 children (89%) in Miami, Florida and 208 of 217 children (96%) in Washington, DC were African-American.

The medical progress made in the treatment of HIV infection with highly active antiretroviral therapies (HAART) has led to a dramatic decline in the incidence of death among adults with HIV-infection. By 1999, however, HIV became the third leading cause of end-stage renal disease (ESRD) among African-Americans aged 20 to 64 years. In contrast to the declining incidence of HIV-infection in the adult population, the incidence of ESRD due to HIVAN has decreased much slower for unknown reasons. The incidence of pediatric AIDS cases also has been declining over the past decade, from 952 new cases diagnosed in 1992 to only 101 in 2001. The impact of the declining incidence of pediatric AIDS cases upon the incidence of pediatric HIVAN remains unknown. The progression of pediatric HIVAN appears to occur more slowly than the adult HIVAN population, with a mean time from initial diagnosis of HIVAN to ESRD of 8 to 20 months. Mortality is high in the pediatric HIV-infected population, with nearly 80% of pediatric patients with HIVAN dying.

For this study, we seek to estimate the prevalence of CKD in HIV-infected patients overall and within specific racial groups.

Participants will be screened with a first-morning macroscopic urinalysis for the detection of proteinuria, and a semi-quantitative measurement of proteinuria using urine protein-to-creatinine and urine microalbumin-to-creatinine ratios. Those patients who have proteinuria of greater than or equal to 1+ on a first-morning macrourinalysis, or a urine protein-to-creatinine ratio of > 0.20 or a urine microalbumin-to-creatinine ratio of > 30 mcg/mg of creatinine, will have a repeat first-morning macroscopic urinalysis, and urine protein-to-creatinine and urine microalbumin-to-creatinine ratios performed 3 months later. Prior to the obtaining of any of the urine samples, those participants who are taking angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) therapy for their anti-proteinuric or anti-hypertensive effects will discontinue their medication for 2 weeks prior to the urine sample collection. After collecting the first-morning urine sample, the study participant may resume his/her prior ACEI or ARB at the previously prescribed dose and schedule. Those patients who have fixed proteinuria on a first-morning macroscopic urinalysis on 2 occasions separated by 3 months will be referred to the Pediatric Nephrology Clinic for further evaluation for proteinuria and/or CKD. The calculated GFR will be determined using the most recent serum creatinine and patient height from the medical record using the Schwartz formula. Chronic Kidney Disease will be defined, as in the NKF KDOQI guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Known/confirmed HIV-infection or AIDS
* Age > 1 but < 21 years of age
* Able to tolerate discontinuation of ACEI or ARB
* Either gender

Exclusion Criteria:

* HIV negative status
* Age < 1 or > 21 years of age
* Unable to tolerate discontinuation of ACEI or ARB

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 320 (Estimated)
Dates: Start 2004-09; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D. McBryde, MD, Principal Investigator — Children's National Research Institute; Susan L. Furth, MD, PhD, Study Director — Johns Hopkins University
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States